CLINICAL TRIAL: NCT01564264
Title: Prospective Cohort Study Evaluating Identification Rate of Sentinel Node in the Management of Endometrial Cancer Utilizing a Combined Method of Cervical and Myometrial Injections
Brief Title: Sentinel Node Biopsy in Endometrial Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hamilton Health Sciences Corporation (Other)
Collaborators: Juravinski Cancer Centre Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SNEndometrialCa
Record Dates: First submitted 2012-03-23; First posted 2012-03-27 (Estimated); Last update posted 2014-09-03 (Estimated); Status verified 2014-08

CONDITIONS: Uterine Neoplasms; Sentinel Lymph Node Biopsy
Keywords: Uterine Neoplasms; Sentinel Lymph Node Biopsy
MeSH Terms: conditions — Uterine Neoplasms | interventions — Sentinel Lymph Node Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sentinel Node Biopsy (Experimental): Each participant will have both measurements, the new diagnostic test (sentinel node biopsy) and the gold standard (complete lymphadenectomy)
  Interventions: Procedure: Sentinel Lymph Node Biopsy

INTERVENTIONS:
Procedure: Sentinel Lymph Node Biopsy — Sentinel node biopsy after injections of 0.4 mci of Technetium 99 in the cervix and 4 mL of Patent Blue into the myometrium followed by standard retroperitoneal lymph node dissection

SUMMARY:
The purpose of this study is to determine if there is a difference between the lymphatic drainage of the cervix and corpus of the uterus after injecting a radiocolloid in the cervix and blue dye in the corpus of the uterus and to investigate the identification rate of sentinel nodes using this technique in patients with cancer of the uterus.

DETAILED DESCRIPTION:
About 20 percent of women diagnosed with uterine cancer have spread outside of the uterus, mainly to the lymph nodes. If these metastases are recognized these women can still be cured with chemotherapy and radiation. Unfortunately different kind of imaging are not very sensitive in identifying patients with lymph node metastases and currently a complete removal of the lymph nodes in the pelvis and around the aorta is the gold standard diagnostic test. Sentinel node biopsy (SLNB) is a surgical technique that aims to identify the nodes that drain specifically the area were the tumor is located. A tracer is injected around the tumor and then the locoregional lymph nodes are tested for the presence of this tracer (blue dye and a radioactive substance). If the sentinel lymph node does not contain cancer, then there is a high likelihood that the cancer has not spread to any other area of the body.The benefits of doing sentinel node biopsy is that it decreases the potential complications associated with the removal of all the lymph nodes. This technique is the standard treatment for other cancers as breast cancer and melanoma and is emerging as a promising technique in gynecological cancers.

There is no agreement regarding the best technique to do SLNB in women with uterine cancer and this procedure is still at the stage of determining feasibility. Since 1996, there have been publications aiming to determine the most appropriate way to do sentinel node in uterine cancer. As the uterus cannot be reached preoperatively for tracer injection, the standard approach for other tumor sites of preoperative peritumoral injection of Technetium 99 followed by intraoperative injection of blue dye has needed to be modified. Blue dye with or without a radiocolloid have been administered either subserously (the uterus outer layer), cervically, dually, and hysteroscopically with a wide range of results in terms of identification rates of sentinel nodes. Certain factors as site of injection, volume and number of injections, interval time since injection to identification of sentinel nodes and surgical approach as laparotomy versus laparoscopy have been associated with the likelihood of identifying these nodes.

This study plans to determine the pattern of lymphatic drainage for the cervix and corpus of the uterus by injecting a different tracer in these 2 sites and also to incorporate all factors that have been proved to be associated with a better identification rate of sentinel nodes in a protocol in order to determine if this technique is feasible and reliable.

ELIGIBILITY:
Inclusion Criteria:

1. Women older than 18 years old
2. Endometrial cancer
3. Histologies: Grade 2 and 3 endometrioid adenocarcinoma, clear cell and papillary serous carcinoma
4. Suitable candidates for surgery
5. Clinically stage 1 or confined to the uterus

Exclusion Criteria:

1. Grade 1 endometrioid adenocarcinoma
2. Metastatic disease

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2012-11; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Location of Sentinel node | Measurement for each participant will be performed between 2-4 hours after injecting Technetium 99 in the cervix
  Locations: internal iliac, external iliac, common iliac, paraaortic or presacral areas Location will be registered by type of sentinel nodes: blue nodes, reflecting the uterine pattern of lymphatic flow (after myometrial injection of blue dye)and hot nodes, reflecting cervical pattern of lymphatic flow (after injection of Technetium 99 in the cervix)

SECONDARY OUTCOMES:
Identification of metastatic lymph nodes by the sentinel node procedure | Measurement will be performed 2-4 hours after the cervical injection with Technetium 99
  Every participant will have a sentinel node procedure followed by a complete removal of the lymph nodes (gold standard), during the same surgery. Accuracy parameters of the sentinel node technique will be compared to the gold standard (complete lymphadenectomy)

CONTACTS AND LOCATIONS:
Overall Officials: Waldo G Jimenez, MD MSc, Principal Investigator — McMaster University
Locations (1):
- Juravinski Hospital, Juravinski Cancer Centre, McMaster University, Hamilton, Ontario, Canada